CLINICAL TRIAL: NCT00138307
Title: Immunological Correlates of Protection Against Clinical Malaria in a Cohort of Young Children in the Kassena Nankana District of Ghana
Brief Title: Correlates of Protection in Ghana
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 04-027
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2007-03

CONDITIONS: Malaria
Keywords: malaria, children, naturally acquired immunity, Ghana
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Malaria is a sickness passed from one person to the other by the bite of a mosquito. In areas of frequent malaria infection, children may develop natural protection against malaria and they are less likely to become sick or die from it as they age. The purpose of this study is to investigate the body's natural protection against malaria in children by testing their blood. This information may help investigators develop a malaria vaccine. The Navrongo Health Research Centre is conducting this study in Ghana. Three hundred healthy children between the ages of 1 and 5 years will participate in the study for 12 months. Study procedures will include 7 field worker visits to check on the child's health and obtain a blood sample. Every two months, a blood sample will be taken from each child to test it for strength against malaria. Whenever a child is sick, the child will be tested for malaria.

DETAILED DESCRIPTION:
The principal aim of this study is to identify immunological correlates of naturally acquired immunity to malaria in young children in the process of acquiring clinical immunity. As a secondary aim, the investigators will study whether allele specific immune responses provide only allele-specific protection against symptomatic infection. Finally, the investigators will assess the baseline immune responses and the extent to which they are boosted during the malaria transmission season in a population likely to be involved in malaria vaccine trials in the near future. The overall study design is to enroll 300 healthy children, aged 1-5 years, located in the northern section of the Kassena-Nankana district and to follow them for twelve months, including the entire high malaria transmission season. They will be evaluated upon enrollment, bimonthly, and at the close of the study by physical examination, malaria smear, hemoglobin determination, and analysis of levels of specific antibody directed against a panel of candidate malaria vaccine antigens. Throughout the course of the study the children will be followed with passive case detection. In between the scheduled visits, parents will be encouraged to bring their children to the Paga Health Centre or Navrongo War Memorial Hospital or to a field worker anytime that they believe the child is not well. At such visits, the child will be evaluated with a morbidity questionnaire including a physical examination. A blood smear will be taken and a rapid malaria diagnostic test (DiaMed Optimal Rapid Malaria test) and hemoglobin measurement will be performed at the time of the visit. Treatment decisions will be based on clinical assessment and the result of the rapid malaria test. The smear result will not be available at the time initial treatment decisions are made. Children diagnosed with malaria will be treated with standard therapy per Ghana Ministry of Health policy by Ghana Health Service personnel. Children suffering from severe anemia or from any form of severe malaria will be referred to the Navrongo War Memorial Hospital for definitive treatment, including intravenous anti-malarial therapy and transfusion, if indicated, at no cost to the subject. At the time of discharge the subject will be evaluated by a study physician with a history and physical, malaria smear and hemoglobin determination. If in the clinical judgment of the study physician no further treatment is required, the subject will resume participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female children aged between 1-5 years.
2. Willingness of parent or guardian to give and sign a consent form and have the child participate in this study.
3. The expectation of continuous residency in the Kassena-Nankana District for the entire study period

Exclusion Criteria:

1. Pre-existing chronic disease at the time of enrollment.
2. Acute illness at the time of enrollment.
3. Hemoglobin less than 6.0g/dL at the time of enrollment.
4. Inability of the child's parent or guardian to give informed consent.
5. Expectation of possible unavailability to continue participation in the study.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300
Dates: Study Completion 2006-03

CONTACTS AND LOCATIONS:
Locations (2):
- Ghana (2):
  - Noguchi Memorial Institute of Medical Research, Legon
  - Navrongo Health Research Centre, Navrongo